CLINICAL TRIAL: NCT04509076
Title: PrEP iT!: A Pilot Test of a Mobile Peer Support Intervention to Optimize PrEP Adherence and Retention in PrEP Care
Brief Title: PrEP iT! Mobile App Intervention
Acronym: PrEP iT!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Hennepin Healthcare Research Institute (Other)
Responsible Party: Principal Investigator, Keith Horvath, Associate Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-2019-0291; R34MH116878 (NIH)
Record Dates: First submitted 2020-03-23; First posted 2020-08-11 (Actual); Results first posted 2023-06-15 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Treatment Adherence and Compliance
Keywords: Pre-Exposure Prophylaxis (PrEP; HIV Prevention
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: 2-arm RCT with 1:1 randomization to PrEP iT! group or the usual care control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PrEP iT! (plus usual PrEP care) (Experimental): The PrEP iT! intervention is a mobile-optimized website with components tailored for young men who have sex with men on PrEP.
  Interventions: Behavioral: PrEP iT! (plus usual PrEP care)
- Usual PrEP care only (Placebo Comparator): Clinic visits every 3 months in the initial period following PrEP initiation, including HIV/STI screening and laboratory toxicity testing
  Interventions: Behavioral: Usual PrEP care

INTERVENTIONS:
Behavioral: PrEP iT! (plus usual PrEP care) — The PrEP iT! intervention is a mobile-optimized website, with the following components:
  * PrEP Adherence, PrEP Appointment, and Sexual Activity Self-Monitoring
  * Tailored feedback on PrEP adherence/non-adherence
  * PrEP and sexual health information tailored for YMSM
  * Text message reminders for PrEP adherence and healthcare appointments
  * An "ask the expert" feature
  Arms: PrEP iT! (plus usual PrEP care)
Behavioral: Usual PrEP care — Clinic visits every 3 months in the initial period following PrEP initiation, including HIV/STI screening and laboratory toxicity testing
  Arms: Usual PrEP care only

SUMMARY:
The long-term goal of this research is to create an effective and sustainable program to support retention in PrEP care and PrEP adherence among 18-29 year old men who have sex with men (MSM). To reach this goal, we will develop and pilot test a mobile intervention tailored to young MSM, called PrEP iT! Primary aims include:

Aim 1: Develop the PrEP iT! mobile intervention through focus groups with young MSM and refine iterations through input from a community advisory board (CAB).

Aim 2: Conduct a pilot randomized controlled trial to assess the feasibility, acceptability and preliminary impact of the PrEP iT! intervention for young MSM.

DETAILED DESCRIPTION:
Study Design:

We propose to evaluate the feasibility, acceptability and preliminary impact of PrEP iT! in a pilot RCT (n=80). Young men who have sex with men (YMSM) recently (re)initiating PrEP will be randomized to receive either PrEP iT! plus usual care or usual care alone, and followed for 6 months with assessments at baseline, and 3- and 6-months.

PrEP iT! will use open source software that conforms to current programming standards, and can be used across all devices (desktop, laptop, smartphone, and tablet) to ensure sustainability. PrEP iT! will be developed from feedback from PrEP-using YMSM through focus groups and a community advisory board (CAB). PrEP iT! is grounded in the Information, Motivation, and Behavioral Skills model, and also draws from a model of technology adoption.

PrEP iT! intervention components are:

* PrEP Adherence, PrEP Appointment, and Sexual Activity Self-Monitoring
* Tailored feedback on PrEP adherence/non-adherence
* PrEP and sexual health information tailored for YMSM
* Text message reminders for PrEP adherence and healthcare appointments
* An "ask the expert" feature

Control arm participants will receive usual PrEP care only. Locally this entails, clinic visits every 3 months in the initial period following PrEP initiation, including HIV/STI screening and laboratory toxicity testing.

Study Sample:

Recruitment will be stratified by age in a 1:1 ratio (i.e., n=40 per group) of 18-24 and 25-29 year olds, and will reflect 50% Black and/or Hispanic YMSM participation. This will allow us to explore subgroup differences (e.g., by age and race/ethnicity) for PrEP iT! to better inform future trials.

Recruitment and Clinical Sites:

Participants will be recruited from two clinics in Minneapolis that provide PrEP care. The clinical sites include the HIV clinic at Hennepin Healthcare (HH) and the Hennepin County STD clinic. We will recruit and enroll study participants concurrent with their PrEP clinical visits when possible.

Participants will be recruited in four ways: a) PrEP clinic patients who are new or returning to care (i.e., are not currently receiving PrEP) will be identified by clinic staff and referred to research coordinators on the day of their clinic visit when possible; b) flyers will be hung in PrEP clinics and other HIV/AIDS NGO service organizations within the Twin Cities; and c) the study team will engage and solicit referrals from other community HIV/AIDS NGO with focused PrEP and prevention campaigns.

Enrollment, Randomization, and Follow-up Visits:

Study candidates will undergo a separate screening visit with a brief questionnaire at/after PrEP clinic visits. Participants will have a rapid HIV test as part of usual care. Persons whose test positive for HIV will be referred for same-day evaluation and care. Participants are randomized 1:1 to either the intervention (PrEP iT! + usual care) or control (usual care) arm. The randomization sequence will be stratified by age (18-24 v. 25-29 yrs) and use blocks of ten.

After informed consent, participants will complete a computer-assisted baseline survey. All participants will be provided usual PrEP educational information encouraged to attend their regular healthcare visits. Participants randomized to the treatment arm (PrEP iT! + usual care) will be guided through setting up their user account and user profile, provided with basic training on how to navigate and use intervention components, and given the opportunity to ask questions. YMSM in the treatment arm will have immediate access to PrEP iT! after the initial visit.

YMSM will undergo a 3- and 6-month follow-up assessment, with multiple reminders sent to participants prior to each visit. The 3- and 6-month stud procedures include completing a short computerized assessment, and submitting a dried blood spot specimen for the TFV-DP analyses. Study data will also be collected from the month 3 and month 6 healthcare visits that include laboratory and clinical data generated routinely as part of standard PrEP care (e.g., testing for HIV Ab and other STIs). We anticipate that most HIV tests results data will be extracted from participant's medical record to confirm their HIV-negative status. In the event that we must conduct an HIV test (e.g., we are unable to extract that from the medical record or if there is an expressed concern that the participant's HIV status has changed), they will be conducted at the Hennepin Healthcare clinical laboratory, using standard clinical assays (we use the HIV Ab/Ag combination test for diagnosis). This information would be captured in our CRFs via REDCap, and this information will be securely transferred to SDSU but would be via a de-identified file.

Study retention protocols involve the use of multiple contact methods, including telephone calls, text messages and e-mail reminders. We anticipate no more than 20% attrition.

Exit Interviews: A random subset of participants randomized to the PrEP iT! arm will be asked if he would be willing to participate in 30-60 minute exit interview to assess a) his experience in the intervention, b) suggestions for modifications to the existing interface, c) suggestions for new features; and d) and changes to the study procedures. Recruitment for exit interviews will entail sufficient numbers for the goal of achieving ten men completing the exit interview.

ELIGIBILITY:
Inclusion criteria for the pilot RCT are:

1. Prescribed PrEP by a healthcare provider;
2. Self-reported 18-29 years of age;
3. Assigned male at birth;
4. Current male gender identification;
5. Gay, bisexual or other non-heterosexual identity or has had sex with a man in the past year;
6. Confirmed HIV-negative status (before starting PrEP);
7. Started PrEP in the past 6 months (either taking PrEP for the first time or restarting PrEP after prior use) and has a current PrEP prescription;
8. English-speaking (as the intervention will be built in English);
9. Able to meet with project staff at baseline and follow-up visits;
10. Regular access to SMS or the internet, either through a mobile device, tablet computer, and/or desktop or laptop computer

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male at birth; Current male gender identification
Enrollment: 80 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-04-15 (Actual); Study Completion 2022-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hennepin County Medical Center, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Horvath KJ, Helm JL, Black A, Chase GE, Ma J, Klaphake J, Garcia-Myers K, Anderson PL, Baker JV. A Pilot Randomized Controlled Trial of an mHealth Intervention to Improve PrEP Adherence Among Young Sexual Minority Men. AIDS Behav. 2024 Aug;28(8):2804-2820. doi: 10.1007/s10461-024-04374-3. Epub 2024 May 31. PMID 38816592

RESULTS

PARTICIPANT FLOW:
Groups:
- PrEP iT! (Plus Usual PrEP Care): The PrEP iT! intervention is a mobile-optimized website with components tailored for young men who have sex with men on PrEP.
  PrEP iT! (plus usual PrEP care): The PrEP iT! intervention is a mobile-optimized website, with the following components:
  * PrEP Adherence, PrEP Appointment, and Sexual Activity Self-Monitoring
  * Tailored feedback on PrEP adherence/non-adherence
  * PrEP and sexual health information tailored for YMSM
  * Text message reminders for PrEP adherence and healthcare appointments
  * An "ask the expert" feature
Period: Overall Study
Arm/Group | PrEP iT! (Plus Usual PrEP Care) | Usual PrEP Care Only
Started | 40 | 40
Completed | 38 | 36
Not Completed | 2 | 4
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PrEP iT! (Plus Usual PrEP Care) | Usual PrEP Care Only | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (2.70) | 25.3 (2.62) | 25.1 (2.65)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 39 | 39 | 78
  Gender nonbinary | 1 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 9 | 18
  Not Hispanic or Latino | 31 | 31 | 62
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 8 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 6 | 13
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: High Protective Level of PrEP Adherence From Tenofovir Diphosphate (TVF-DP) Levels
Description: Adherence thresholds estimated through analysis of tenofovir diphosphate (TVF-DP) levels from dried blood spot (DBS) specimens were used to categorize each participant as having a high protective level (i.e., a high likelihood of protection from HIV) of PrEP (800 or greater of emtricitabine-tenofovir disoproxil fumarate [FTC-TDF] and 950 or greater of FTC-tenofovir alafenamide [FTC-TAF]) or not. Results reported here are for high protective levels of PrEP.
Time Frame: 6-month follow up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP iT! (Plus Usual PrEP Care) | Usual PrEP Care Only
Number analyzed (Participants) | 27 | 24
Participants | 13 | 15

2. Primary Outcome: Proportion of Participants With High Self-reported PrEP Adherence in the Past 7 Days
Description: Participants were asked at the month 6 survey to respond to the following item: "In the past 7 days, how many days did you take PrEP?" Response options ranging from 0 days to 7 days, with 1 day increments. Responses of 4, 5, 6, or 7 days were categorized as having a high protective level of PrEP (i.e., a high likelihood of protection from HIV). Results reported here are for high protective levels of PrEP.
Time Frame: 6-month follow up assessment
Measure: Count of Participants; unit: Participants
Arm/Group | PrEP iT! (Plus Usual PrEP Care) | Usual PrEP Care Only
Number analyzed (Participants) | 38 | 35
Participants | 27 | 22

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for a period of 9 months.
Arm/Group | PrEP iT! (Plus Usual PrEP Care) | Usual PrEP Care Only
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

LIMITATIONS AND CAVEATS:
This study was designed and conducted as a pilot trial. The goal was to initially evaluate the PrEP-iT! intervention strategy and inform the development of larger definitive clinical trial. Thus, power was limited for outcome comparisons and future larger trials are needed to formally assess efficacy of the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-14): https://cdn.clinicaltrials.gov/large-docs/76/NCT04509076/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-19): https://cdn.clinicaltrials.gov/large-docs/76/NCT04509076/ICF_001.pdf